CLINICAL TRIAL: NCT03012529
Title: CSP #2001 - Investigation of Rifampin to Reduce Pedal Amputations for Osteomyelitis in Diabetics (VA Intrepid)
Brief Title: Investigation of Rifampin to Reduce Pedal Amputations for Osteomyelitis in Diabetics
Acronym: VA INTREPID
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2001
Record Dates: First submitted 2016-12-22; First posted 2017-01-06 (Estimated); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Osteomyelitis; Diabetes; Amputation
Keywords: Rifampin; Double-blind; Clinical Trial; Veterans; Diabetes
MeSH Terms: conditions — Osteomyelitis; Diabetes Mellitus | interventions — Rifampin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active drug (Active Comparator): Patients receive oral adjunctive rifampin therapy
  Interventions: Drug: Rifampin
- Placebo (Placebo Comparator): Patients receive oral riboflavin
  Interventions: Drug: Riboflavin Placebo

INTERVENTIONS:
Drug: Rifampin — Subjects who are randomly assigned to adjunctive rifampin will receive a 600 mg oral daily dose targeted for a six-week period. If a subject experiences gastrointestinal intolerance on once daily dosing, the study drug may be administered as rifampin 300 mg twice a day.
  Arms: Active drug
Drug: Riboflavin Placebo — A placebo capsule will be administered daily to match frequency and duration of rifampin interventional drug. For the purpose of mimicking urine discoloration when taking rifampin, riboflavin will be added to the placebo to produce a urine discoloration effect.
  Arms: Placebo

SUMMARY:
The purpose of this research study is to determine if rifampin, an antibiotic (a medicine that treats infections), is effective in treating osteomyelitis (infection of the bone) of the foot in diabetic patients. Despite use of powerful antibiotics prescribed over a long period of time, many diabetic patients remain at a high risk for needing an amputation of part of the foot or lower leg because the osteomyelitis is not cured. Some small research studies have shown that addition of rifampin to other antibiotics is effective in treating osteomyelitis in both diabetics and non-diabetics. However, because few diabetics with osteomyelitis have been studied, there is no definite proof that it is better than the usual treatments for diabetic patients. If this study finds that adding rifampin to the usual antibiotics prescribed for osteomyelitis reduces the risk for amputations, doctors will be able to more effectively treat many Veteran patients with this serious infection. Improving treatment outcomes is an important healthcare goal of the VA.

DETAILED DESCRIPTION:
This is a prospective, randomized, double-blind, placebo-controlled, investigation of a six week course of adjunctive rifampin vs. adjunctive matched placebo (riboflavin) added to backbone antibacterial therapy for the treatment of diabetic foot osteomyelitis. Backbone antibacterial therapy will be with single or multiple agents selected by the clinical treatment team based either on culture results or standard empiric therapy, and which can be administered either intravenously or orally. Rifampin will be dosed at 600 mg daily. The primary outcome measure is amputation-free survival. Amputation events include both below- and above-ankle amputations. Primary outcomes will be determined by systematic medical record review and through confirmatory research visits, phone calls and, as needed, information from non-VA providers. The results for amputation-free survival will be analyzed by means of a two-sided log-rank test. The secondary outcomes of complete wound epithelialization and remission of osteomyelitis will be determined by the research team through VA record review and/or direct examination.

The study will initially enroll and randomize a total of 880 study participants to receive either rifampin or placebo (riboflavin) in addition to backbone antibiotic therapy prescribed by their clinician. Investigators expect to enroll, on average, close to one subject per month per site (10-12 per year/site) at 28 VA medical centers to achieve total randomization of 880 subjects over seven years. In meeting this average site enrollment projection, Investigators anticipate variation in enrollment between larger and smaller sites, and between high-performing and low-performing sites. Subjects will be followed through the end of the second year after randomization or until a study primary endpoint event (amputation or death) occurs. On average, study participants will be followed for 1.8 years through systematic review of medical records, and by study visits and phone calls.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 and 89 years
2. Diagnosis of diabetes mellitus, either by: 1) use of oral hypoglycemic agents or insulin at the time of enrollment; 2) a hemoglobin A1c (HgA1c) level within the past 90 days > 6.5; or 3) a medical record diagnosis of diabetes mellitus by a clinician on two or more occasions in the previous 10 years
3. Definite or probable osteomyelitis in the diabetic foot, as defined by the International Working Group on the Diabetic Foot (Table 1). Criteria must be present at some point within 90 days prior to enrollment.
4. All planned debridement has been completed prior to randomization.
5. A course of backbone antimicrobial therapy has been selected.

Exclusion Criteria:

1. Patient unable to receive enteral medication.
2. Patient is allergic to or intolerant of rifampin.
3. Patient is taking a drug that has interactions with rifampin that would require either stoppage, substitution or an empiric dose modification that may place the patient at medical risk.
4. Within 30 days of enrollment, patient is taking immunosuppressive medications to prevent rejection of an organ transplant or is receiving chemotherapy for cancer or molecularly targeted therapies for cancer.
5. Patient is receiving antiretroviral therapy for HIV or antiviral medication for Hepatitis C.
6. Patient is participating in another interventional clinical trial for which a waiver of dual enrollment with CSP#2001 has not been obtained.
7. Patient has an ALT > 3 times the upper limit of normal for the site laboratory, or total bilirubin > 2.5 times the upper limit of normal for the site laboratory*,***; INR > 1.5, OR patient has Child-Pugh Class C Cirrhosis.
8. Patient has a baseline white blood cell count (WBC) <2000 cells/mm3*** OR absolute neutrophil count (ANC) <1000 cells/mm3*** OR platelet count <50,000 cells/mm3**,*** OR hemoglobin <8.0 g/dL.**,***.
9. Women of child-bearing potential (those with menses within the last year) with a positive serum pregnancy test.
10. Patient is believed unlikely to be able to complete the trial due to medical conditions.
11. Patient is believed unlikely to complete the trial due to neurologic and psycho-behavioral disorders such as active substance abuse or dependence, disabling dementias or psychoses.
12. Patient refuses or is clinically unable to undergo the recommended level of debridement.
13. Indwelling hardware present in the foot, at the site of the index osteomyelitis.
14. Treatment with antibacterial agents for infection at another site, where the duration of treatment is anticipated to be greater than 14 days.
15. Patient is receiving therapy for COVID-19 that interacts with rifampin.

    * Patients with total bilirubin > 2 times the ULN who have Gilbert's Disease or any other inherited disease affecting bilirubin metabolism without meeting other exclusionary criteria, may be considered for inclusion in the study.

      * Patients with platelet count <50,000 cells/mm3 due only to hypersplenism and meeting no other exclusionary criteria may be considered for inclusion in the study.

        * If multiple laboratory values are available, the most recent value will be applied for eligibility.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 843 (Actual)
Dates: Start 2018-01-22 (Actual); Primary Completion 2025-11-05 (Actual); Study Completion 2025-11-05 (Actual)

PRIMARY OUTCOMES:
Amputation-Free Survival | Assessed 2 years post intervention
  The primary endpoint is amputation-free survival, ending with amputation or death from any cause. Amputation is defined as surgical treatment of osteomyelitis by removal or debridement of necrotic/infected bone (all or part of a bone) from a lower extremity limb or digit on the ipsilateral side of the protocol-treated osteomyelitis. Debridement prior to randomization may include removal of bone. Because this debridement occurs early, prior to exposure to study drug or placebo, removal of bone at that time is not a study endpoint.

SECONDARY OUTCOMES:
Time to Amputation | Assessed 2 years post intervention
  Time from randomization to the occurrence of the components of the primary outcome:
  1. the first occurrence of ipsilateral amputation alone
  2. the first occurrence of ipsilateral above-ankle amputation
  3. the first occurrence of ipsilateral through the ankle (e.g. Symes amputation) or below-ankle amputation proximal to the metatarsal-phalangeal joint
  4. the first occurrence of ipsilateral below-ankle amputation at or distal to the metatarsal-phalangeal joint
  5. all cause death
  Endpoint will be determined by chart review by the Study Coordinator, with confirmation by the Site Investigator, and as needed, by the Study Chair.
New course of antibacterial therapy for ipsilateral foot infection | Assessed 2 years post intervention
  New courses of antibacterial therapy for ipsilateral foot infection during the first year after randomization (yes/no per patient).
  Endpoint will be determined by chart review by the Study Coordinator, with consultation with the Site Investigator as needed to confirm that the new course of treatment is directed toward continued or recurrent osteomyelitis of the initially affected lower extremity. The new course will require there be at least a 14 day interval between the end of the initial back-bone antibiotic therapy course.
Quality of Life - SF-36 | Assessed 12 months post intervention
  Quality of life, measured by the 36-Item Short Form Health Survey (SF-36; Ware & Sherbourne, 1992) and its physical and mental health subscales.
  This is a widely used self-report instrument that will be administered by the Study Coordinator at baseline, 3-, 6- and 12-months.
Ambulatory Status | Assessed 12 months post intervention
  Ambulatory status, measured by the Study Coordinator, using a modified item from the Amputee Mobility Predictor Questionnaire56.
  The patient's "usual method of ambulation within the home" will be assessed by a single self-report item at baseline, 3-, 6- and 12-months using the following response categories:
  1. No assistive device required to move about
  2. Cane
  3. Crutches
  4. Walker
  5. Wheelchair
  6. Bed bound
Incidence of Falls | Assessed 12 months post intervention
  Incidence of falls, measured by self-reported frequency of falls and falls that required medical attention in the one-month periods preceding research visits at Baseline, 3-, 6- and 12-months.
Incidence of adverse events related to direct toxicity of rifampin | Assessed 3 months post intervention
  Incidence of adverse events related to direct toxicity of rifampin in active drug vs. placebo groups:
  1. Nausea requiring dividing the dose to twice a day
  2. Rash requiring study drug discontinuation
  3. Nausea requiring study drug discontinuation
  4. Grade 3 or 4 liver enzyme (ALT) elevations Local Site Investigators, with assistance from their Study Coordinators, will be responsible for reporting adverse events which will be used to analyze these secondary endpoints.
Incidence of adverse events from drug interactions | Assessed 3 months post intervention
  Incidence of adverse events from drug interactions in active drug vs. placebo groups:
  1. Cardiovascular: Myocardial infarction, cerebrovascular accident, hospitalization for hypertensive emergency
  2. Glycemic control: Hospitalization for a primary diagnosis of hypoglycemia or uncontrolled diabetes Local Site Investigators, with assistance from their Study Coordinators, will be responsible for reporting adverse events which will be used to analyze these secondary endpoints.
Comparative dropout | Assessed 6 weeks post intervention
  Overall comparative dropout data during the 6-week intervention based on drug intolerance/drug interactions/adverse events in active drug vs. placebo groups.
  Dropout endpoint will be determined by chart review by the Study Coordinator and by telephone calls to the subject.
Remission of osteomyelitis | Assessed at 1 year post intervention
  Remission of osteomyelitis at 12 months (yes/no). Remission is defined as epithelialization of any overlying soft tissue defect and the absence of local signs and symptoms of inflammation.
  Endpoint will be determined by physical examination by the Site Investigator at the 12 month visit.
Complete epithelialization of the wound | Assessed 1 year post intervention
  Complete epithelialization of the wound at 6 weeks and at 3, 6 and 12 months (yes/no).
  Endpoint will be determined by physical examination by the Site Investigator at the 3, 6 and 12 month visits.
First occurrence of ipsilateral amputation related to index osteomyelitis | Assessed 2 years post intervention
  Time from randomization to the first occurrence of ipsilateral amputation for the treatment of osteomyelitis related to the index osteomyelitis.
  Relatedness will be determined by the LSI or qualified Co-investigator on thePrimary Outcome case report form. An episode of ipsilateral osteomyelitis is considered related to the index osteomyelitis if it involves the same bone or a contiguous bone.

CONTACTS AND LOCATIONS:
Overall Officials: Mary T Bessesen, MD, Study Chair — Rocky Mountain Regional VA Medical Center, Aurora, CO
Locations (30):
- United States (30):
  - Phoenix VA Health Care System, Phoenix, AZ, Phoenix, Arizona
  - VA Loma Linda Healthcare System, Loma Linda, CA, Loma Linda, California
  - VA Long Beach Healthcare System, Long Beach, CA, Long Beach, California
  - VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California
  - VA Northern California Health Care System, Mather, CA, Sacramento, California
  - VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California
  - Rocky Mountain Regional VA Medical Center, Aurora, CO, Aurora, Colorado
  - Washington DC VA Medical Center, Washington, DC, Washington D.C., District of Columbia
  - Bay Pines VA Healthcare System, Pay Pines, FL, Bay Pines, Florida
  - North Florida/South Georgia Veterans Health System, Gainesville, FL, Gainesville, Florida
  - Miami VA Healthcare System, Miami, FL, Miami, Florida
  - James A. Haley Veterans' Hospital, Tampa, FL, Tampa, Florida
  - Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia
  - VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan
  - Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota
  - St. Louis VA Medical Center John Cochran Division, St. Louis, MO, St Louis, Missouri
  - James J. Peters VA Medical Center, Bronx, NY, The Bronx, New York
  - Salisbury W.G. (Bill) Hefner VA Medical Center, Salisbury, NC, Salisbury, North Carolina
  - Cincinnati VA Medical Center, Cincinnati, OH, Cincinnati, Ohio
  - Louis Stokes VA Medical Center, Cleveland, OH, Cleveland, Ohio
  - Dayton VA Medical Center, Dayton, OH, Dayton, Ohio
  - Oklahoma City VA Medical Center, Oklahoma City, OK, Oklahoma City, Oklahoma
  - VA Portland Health Care System, Portland, OR, Portland, Oregon
  - Tennessee Valley Healthcare System Nashville Campus, Nashville, TN, Nashville, Tennessee
  - VA North Texas Health Care System Dallas VA Medical Center, Dallas, TX, Dallas, Texas
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas
  - South Texas Health Care System, San Antonio, TX, San Antonio, Texas
  - VA Salt Lake City Health Care System, Salt Lake City, UT, Salt Lake City, Utah
  - Salem VA Medical Center, Salem, VA, Salem, Virginia
  - William S. Middleton Memorial Veterans Hospital, Madison, WI, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bessesen MT, Doros G, Henrie AM, Harrington KM, Hermos JA, Bonomo RA, Ferguson RE, Huang GD, Brown ST. A multicenter randomized placebo controlled trial of rifampin to reduce pedal amputations for osteomyelitis in veterans with diabetes (VA INTREPID). BMC Infect Dis. 2020 Jan 8;20(1):23. doi: 10.1186/s12879-019-4751-3. PMID 31914940